CLINICAL TRIAL: NCT04900454
Title: A Phase 1 Study of DVX201, an Allogeneic Natural Killer (NK) Cell Therapy in Subjects Hospitalized for COVID-19
Brief Title: Allogeneic Natural Killer (NK) Cell Therapy in Subjects Hospitalized for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coeptis Therapeutics (Industry)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVX201-COV-01; RG1121470 (Other: Fred Hutchinson Cancer Research Center)
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Pneumonia
Keywords: NK cells; Cell therapy; Allogeneic

STUDY DESIGN:
Intervention Model Description: This is an, open-label, non-randomized Phase 1 dose-finding study of DVX201 in patients hospitalized with COVID-19. Subjects will enroll and the MTD and/or the RP2D of DVX201 will be determined utilizing a modified "3+3" enrollment schema.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DVX201 infusion (Experimental): Subjects will enroll and the MTD and/or the recommended phase 2 dose of DVX201 will be determined utilizing a modified "3+3" enrollment schema.
  This study will enroll a minimum 3 subjects who each receive a single dose of DVX201 and who are evaluable for toxicities at each dose level. Depending on the occurrence of DLTs and the number of dose levels evaluated, additional subjects may be enrolled (approximately 3-15 additional subjects). All subjects will be followed for 28 days post infusion of DVX201.
  Interventions: Biological: DVX201

INTERVENTIONS:
Biological: DVX201 — Single infusion of DVX201, an allogeneic NK cell therapy derived from CD34+ hematopoietic stem cells

SUMMARY:
This study is being done to determine the highest tolerated dose of an investigational cell therapy called DVX201 in patients hospitalized with COVID-19. DVX201 is an allogeneic NK (natural killer) cell therapy. NK cells are a normal part of your immune system that have the ability to identify and kill cells in the body that are infected by viruses such as COVID-19. There is evidence that both NK cell exhaustion and low numbers of NK cell in the blood occur in COVID-19 patients, and this may contribute to worsening of the infection. Therefore, infusion of healthy functional NK cells (like DVX201) may help overcome COVID-19 infection and prevent progression of the disease. This study is being done to look at the safety and tolerability of DVX201 in patients with COVID-19 and to gather information on how COVID-19 responds to treatment with DVX201.

ELIGIBILITY:
Inclusion Criteria:

1. Be capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
2. Be between 18 and 80 years of age and weigh at least 40 kg, inclusive, at time of informed consent
3. Be confirmed positive for COVID-19 (SARS-CoV-2) infection as determined by validated clinical PCR assay or by a hospital validated serological test within 7 days of consent
4. Symptomatic onset within 7 days of signing consent
5. Require hospitalization and meet the following:

   1. Radiographic infiltrates by imaging (chest x-ray, CT scans)
   2. Able to maintain a SpO2 ≥ 93% at rest. Supplemental oxygen to a maximum 4L by low flow O2-delivery is allowed, but not required
   3. Meet 2 out of the 3 following criteria:

   i. IL-6 < 150 pg/mL ii. CRP < 100 mg/L (10 mg/dL) iii. Ferritin < 1000 ng/mL
6. Women/men of reproductive potential must have agreed to use an effective contraceptive method during the study and for a minimum of 90 days after study treatment

Exclusion Criteria:

1. Weight less than 40 kg
2. Be ventilator dependent or be diagnosed with ARDS or multi-system organ failure
3. Have elevated oxygen requirement exceeding 4L oxygen by nasal cannula
4. Expected intubation within 24 hours per investigators assessment
5. Expected discharge from hospital within 72 hours of planned DVX201 date of infusion
6. Have a known hypersensitivity to constituents of DVX201, such as DMSO or atinhistamine medications
7. Have a history of symptomatic pulmonary or chronic pulmonary disease or severe asthma on chronic therapy for treatment
8. Have a history of baseline requirement of supplemental oxygen prior to COVID-19 diagnosis
9. Active autoimmune disorder or other medical condition requiring systemic immunosuppressive therapy (including steroids at > 5 mg prednisone or equivalent daily)
10. Be pregnant or breast-feeding
11. Have inadequate organ function as defined by:

    1. Acute or chronic kidney injury requiring intermittent or continuous venovenous hemodialysis or estimated GFR of < 60 mL/min/1.73 m2
    2. Abnormal liver function defined by AST (aspartate aminotransferase), ALT (alanine aminotransferase) or alkaline phosphatase ≥ 5 times the upper limit of normal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLT) | 7 days
  DLTs defined as grade 3 or greater infusion related reactions within 24 hours and any treatment emergent toxicity grade 3 or greater within 7 days apart from known complications of COVID-19

SECONDARY OUTCOMES:
reduction/clearance of viral load/viral shedding | through study completion, an average of 28 days post cell infusion
  time in days to clearance of virus
Oxygen requirements | through study completion, an average of 28 days post cell infusion
  Time in days on supplemental oxygen and time in days to resolution of hypoxia
Disease progression | through study completion, an average of 28 days post cell infusion
  Incidence of disease progression to ICU admission and/or ventilatory support
CRS | through study completion, an average of 28 days post cell infusion
  Incidence of cytokine release syndrome requiring clinical intervention
hospital discharge | through study completion, an average of 28 days post cell infusion
  Time in days post infusion of DVX201 to hospital discharge

OTHER OUTCOMES:
Length of time that DVX201 (NK cells) remain in the blood | through 28 days post infusion
  Evaluation of persistence of DVX201 in the peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Josh Hill, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Medical Center, Seattle, Washington, United States